CLINICAL TRIAL: NCT03577522
Title: Randomized Controlled Trial Comparison of Two Hydroxy-apatite Coated Hip Stems Utilizing Radiostereometric Analysis
Brief Title: Comparison of Two Hydroxy-apatite Coated Hip Stems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B2018-031
Record Dates: First submitted 2018-06-20; First posted 2018-07-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Avenir cementless hip stem (Active Comparator): Total hip arthroplasty: Avenir vs Corail
  Interventions: Device: Avenir cementless hip stem
- Corail HA-coated hip stem (Active Comparator): Total hip arthroplasty: Corail vs Avenir
  Interventions: Device: Corail HA-coated hip stem

INTERVENTIONS:
Device: Avenir cementless hip stem — Avenir cementless hip stem vs Corail HA-coated hip stem
  Arms: Avenir cementless hip stem
Device: Corail HA-coated hip stem — Avenir cementless hip stem vs Corail HA-coated hip stem
  Arms: Corail HA-coated hip stem

SUMMARY:
In this study, the investigators propose to randomize 80 subjects to receive either the Avenir cementless hip stem or a competing, HA-coated hip stem (Corail, DePuy-Synthes) and follow these patients for a period of 2 years post-surgery. The investigators aim to determine if the Avenir cementless hip stem has equivalent or better fixation and clinical outcomes compared to a predicate hip stem with longer clinical history.

DETAILED DESCRIPTION:
This is a multi-center, randomized controlled trial of patients undergoing primary total hip arthroplasty. This study will be focused on enrollment at a single site with possible expansion to additional centers should patient enrollment occur at a slower than expected rate. Decision to expand the study to additional centers will be mutually agreed upon by both the clinical site and the study sponsor.

Patients will be randomized to two study groups:

1. Zimmer Avenir cementless, HA-coated femoral hip stem with matching Trilogy IT cup;
2. DePuy-Synthes Corail cementless, HA-coated, non-collared femoral hip stem with matching Pinnacle cup Patient allocation to the study groups will occur following a randomized 4-block design.

ELIGIBILITY:
Inclusion Criteria

* Symptomatic osteoarthritis of the hip undergoing primary total hip arthroplasty
* Between the ages of 18 and 79 inclusive
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria

* Requires specialty implant (e.g., suspected metal allergy, coxa vera implant)
* Avascular necrosis
* Unresolved infection of the hip
* Hip fracture
* Hip dysplasia
* At risk for loss to follow-up
* Prior surgery to the ipsilateral hip
* Severe proximal femoral deformity preventing the use of standard proximal press-fit femoral components
* Medical condition precluding major surgery
* Current or pending patient incarceration

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Migration | 2 years
  Measured via radiosteriometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Concordia Joint Replacement Group
Locations (1):
- Concordia Hospital, Winnipeg, Manitoba, Canada